CLINICAL TRIAL: NCT06882668
Title: Role of Cardiovascular Imaging in the Early Diagnosis of Hypertrophic Cardiomyopathy in Women
Acronym: IMAGE-HCM
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Azienda Sanitaria Universitaria Giuliano Isontina [ASUGI], Università di Trieste, Italy (Unknown)
Responsible Party: Principal Investigator, Agricola Eustachio, Associate Professor, IRCCS San Raffaele
Other Study IDs: 2022KMEEJF
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Hypertrophic Cardiomyopathy (HCM)
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Hypertrophic cardiomyopathy (HCM) is the most common genetic cardiac disorder worldwide with a prevalence of 1:500 in the general population. It is mainly associated to mutations in genes encoding cardiac sarcomere proteins and it is characterized by left ventricular hypertrophy that is not explained by pathological loading conditions or coexisting myocardial storage disease. In this setting, diagnosis is based on left ventricular wall thickness segment (LVWT) of at least 15 mm documented by echocardiography, cardiac magnetic resonance (CMR) or cardiac computed tomography. Less severe grades of hypertrophy (13-14 mm) are needed when genetic tests are performed and a pathogenic or a likely pathogenic variant documented. However, women with HCM tend to be underdiagnosed or diagnosed at late stages possibly developing unfavorable outcomes. Asymmetry is the hallmark feature of hypertrophy in HCM: rather than by a single segment measurement, the heterogeneity of wall thickness may be better assessed by WTSD, the standard deviation of wall thickness, previously derived in a CMR study.

WTSD with a cut-off of >2.4 had the highest accuracy to identify HCM from normal hearts and from other forms of myocardial hypertrophy in a cohort of living subjects, and was particularly accurate in diagnosing HCM in females.

This is an observational multicentre, prospective study that will explore the combined predictive value of clinical, electrocardiographic and imaging parameters in diagnosing HCM in subjects with clinical suspicion of the disease. Specifically, we will focus on the predictive power of WTSD in diagnosing HCM n women. Indeed, since WTSD with a cut-off > 2.4 to detect HCM was derived from a CMR study, we will test the feasibility of WTSD analysis on echocardiographic imaging and its reliability compared to WTSD analysis on CMR. Exploratory objectives will evaluate the role of WTSD to predict HCM with a cut-off >2.4 also in male population.

This is an observational multicentre, prospective study that will involve 2 Research Units (RU):

* RU1. Cardiovascular Imaging Unit, Hypertrophic Cardiomyopathy Outpatient Clinic, Vita-Salute San Raffaele University/IRCCS San Raffaele Hospital, Milan, Italy.
* RU2. Cardiothoracic and Vascular Department, Heart Failure and Cardiomyopathy Unit, University of Trieste, Azienda Sanitaria Universitaria Giuliano Isontina, Triest, Italy.

The enrolment phase will take up to 18 months (month 1 to 18) (RU1, RU2). Enrolment will prospectively involve:

* All consecutive subjects with suspicion of HCM who are addressed by a general Cardiologist to the 2 RUs for the diagnostic work-up and thus with a high probability of being affected by HCM
* All first-degree relatives of HCM patients already in follow-up at the participating centres.

We consider a proportion of patients who will be classified as dropouts from the study because they will not be diagnosed with HCM.

At time of enrolment (time 0) all patients will be evaluated in ambulatory care setting and will undergo electrocardiogram, transthoracic echocardiography (TTE), CMR and genetic testing.

At 6 month follow-up clinical examination, electrocardiogram and transthoracic echocardiography will be performed in all patients.

The end of enrolment is estimated at 18th month and the follow-up of each patient is estimated at least 6 months. Each patient's clinical, electrocardiographic, and imaging data from the hospital records will be collected. WTSD will be measured both at echocardiography and CMR. All echocardiographic examinations and CMRs will be reviewed and analyzed by a core lab placed at the Cardiovascular Imaging Unit of IRCCS San Raffaele Hospital in Milan, Italy.

ELIGIBILITY:
Inclusion Criteria:

* Able to sign informed consent.
* First-degree relatives of HCM patients already in follow-up at the participating centres, independently from the genetic status of the affected family member.
* Unselected subjects referred to the Cardiomyopathy Outpatient Clinics with clinical suspicion of HCM.
* Availability to perform transthoracic echocardiographic imaging, and to perform CMR.

Exclusion Criteria:

* Known history of systemic hypertension with documented secondary LV heart disease.

  * Known grown up congenital heart disease patients with documented secondary LV hypertrophy.
  * Known hemodynamically relevant valvular diseases with documented secondary LV hypertrophy.
  * Known HCM phenocopies: infiltrative diseases mimicking HCM (cardiac amyloidosis, haemochromatosis and secondary hemosiderosis), metabolic storage diseases (Anderson-Fabry disease, Pompe disease, Danon disease, PRKAG2-related disease).
  * Neuromuscular diseases as Friedreich ataxia, distrophinopathies and desminopathies.
  * Known mitochondrial diseases with documented myocardial involvement.
  * Known malformation syndromes as RAS/MAPK disorders (Noonan syndrome, LEOPARD syndrome, Costello syndrome), cardiofaciocutaneous syndrome.
  * Previous long-term treatment with tacrolimus, hydroxychloroquine, steroids.
  * Known absolute contraindications to CMR.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be composed of all consecutive subjects with suspicion of HCM who are addressed to the 2 Research Units involved by a general Cardiologist for the diagnostic work-up and thus with a high probability of being affected by HCM.
  We consider a proportion of patients who will be classified as dropouts from the study because they will not be diagnosed with hypertrophic cardiomyopathy.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
WTSD | Time point(s) Time 0 Time 6 months
  To validate the feasibility and reliability of WTSD measurements obtained via transthoracic echocardiography (TTE) in women, using a cut-off value of >2.4 mm, by comparing these measurements to WTSD values obtained through cardiac magnetic resonance (CMR) imaging, the established reference standard for WTSD analysis in diagnosing hypertrophic cardiomyopathy (HCM).

CONTACTS AND LOCATIONS:
Locations (1):
- Vita Salute San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided